CLINICAL TRIAL: NCT05599139
Title: The Uptake of Radioactive Iodine Before and After a Low Iodine Diet in Patients With Differentiated Thyroid Carcinoma
Brief Title: Iodine Uptake After a Low Iodine Diet
Acronym: IULID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL65923.042.18
Record Dates: First submitted 2022-10-25; First posted 2022-10-31 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Differentiated Thyroid Cancer
Keywords: Low iodine diet; Iodine uptake

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low iodine diet (Other): Patients recieve a low iodine diet. Consecutive iodine uptake measurements will be made before and after starting this low iodine diet. This study is constructed of only one study arm, and patients will be compared to themselves.
  Interventions: Behavioral: Low iodine diet

INTERVENTIONS:
Behavioral: Low iodine diet — Before ablation and possible subsequent therapy with 131I, patients have to follow a low iodine diet (LID), reducing the iodine intake < 50 mcg per day and thereby depleting the overall iodine store in the body.

SUMMARY:
The goal of this clinical trial is to compare the difference in thyroid uptake of a low dose radioactive iodine (10 MBq 123-I or 37 MBq 123-I) in athyreotic patients with differentiated thyroid carcinoma before and after a low iodine diet (LID) of 7 days.

The main question it aims to answer is:

• What is the difference in iodine uptake before and after a LID of 7 days?

Uptake of a low dose of 123-iodine will be measured in participants before and after a low iodine diet of 7 days. Researchers will compare the uptake (%) before and after the LID.

DETAILED DESCRIPTION:
Rationale:

Differentiated thyroid carcinoma (DTC) is the most common form of thyroid cancer. The initial treatment of DTC consists of a total thyroidectomy followed by ablation therapy with radioactive iodine (131I) which destroy residual thyroid (cancer) tissue. Before starting the (ablation) therapy with 131I, patients have to follow a low iodine diet (LID) reducing the iodine intake < 50 mcg per day. Depleting the overall iodine store in the body theoretically maximizes the expression of the sodium-iodine symporter (NIS). This increased NIS expression results in an increase of the uptake of 131I in remaining thyroid (cancer) cells during 131I therapy and therefore improves the ablation success rates. However, there is no prospective data to support this, merely some retrospective contradictionary data. Patients experience the strict adherence to LID as stressful, distasteful and overwhelming in combination with a new diagnosis of cancer and withdrawal from thyroid hormone. Besides, they are afraid to apply the LID inadequately, which complicates achieving a balanced diet, essential in cancer recovery.

Objective:

To compare the difference in thyroid uptake of a low dose radioactive iodine (10 MBq 123I or 37 MBq 123I), in DTC patients after thyroidectomy, before and after a LID of 7 days.

Study design: observational, single center study performed in the University Medical Center Groningen (UMCG) Groningen, the Netherlands.

Study population: Patients, men and women above the age of 18 years, with a histopathological confirmed diagnosis of DTC who will receive 131I ablation therapy and have to follow a LID according to the Dutch DTC guideline.

Main study parameters/endpoints: The primary endpoint is the clinical relevant difference of a twofold uptake increase, in the thyroid remnant after thyroidectomy in DTC patients, a 10 MBq 123I or 37 MBq 123I tracer dose before and after a LID of 7 days.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

* Burden: Low risk patients (according to the Dutch DTC guideline) will receive 10 MBq 123I twice, followed by a thyroid uptake measurement and will have to collect their urine for 24 hours twice. High risk patients (according to the Dutch DTC guideline) will receive 10 MBq 123I once, followed by a thyroid uptake measurement and have to collect their urine for 24 hours twice. On the day of the first administration of 10 MBq 123I, 1 blood sample (5 ml) will be collected. Low risk patients have to make three additional site visits to the UMCG, high risk patients two additional site visits.
* Risks: The administration of two times 10 MBq will lead to an extra radiation exposure of 0,76 mSv for low risk patients and 0,38 mSv for high risk patients. Blood sampling carriers a negligible risk of a hematoma. The 24 hours urine collection is without additional risk for the patient or the lab technician.

The note of the daily food intake is without additional risk for the patient.

- Benefits: None, participants will participate based on altruistic motives.

ELIGIBILITY:
Inclusion Criteria:

* Patients, men and women above the age of 18 years, have to be diagnosed with DTC and have to follow a LID prior to the 131I ablation therapy according to the Dutch DTC guideline
* Patients have to be fit to adhere to the study protocol
* Patients have to be able to read and understand the Dutch language

Exclusion Criteria:

* Age < 18 years
* Patients using amiodarone
* Patients receiving iodinated contrast < 3 months before the LID
* Pregnancy
* Patients prepared for ablation therapy with rhTSH
* Renal impairment, EGFR <30ml/min/1,73m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Iodine uptake | 7 days
  Difference in iodine uptake in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Zandee, Dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
The IPD will not be available to other researchers as this is not included in the patient consent.